CLINICAL TRIAL: NCT03446950
Title: Candy Cane vs. Boot Stirrups in Vaginal Surgery: A Randomized Control Trial
Brief Title: Study Investigating Role of Unalike Patient Positioning on PROMIS Scores
Acronym: STIRUPPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Sean Francis, Chairperson & Assoc Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 18.0061
Record Dates: First submitted 2018-02-11; First posted 2018-02-27 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Physical Activity; Surgery; Vaginal Hysterectomy; Vaginal Surgery
Keywords: vaginal surgery; patient position; stirrups; functional status; urogynecology
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: To compare patient positioning during vaginal surgery we plan to conduct a single site single blinded randomized controlled trial where patients planning elective vaginal surgery will be randomized to be positioned in Candy cane or Boot stirrups
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to their intervention group. Investigators following up with participants at 6 weeks will be blinded to the group allocation of the participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Candy Cane (Active Comparator): Participants in this arm will be positioned with their legs in candy cane stirrups. Patients will then undergo scheduled vaginal surgery and be asked to complete PROMIS questionnaires before and after surgery.
  Interventions: Procedure: Vaginal Surgery
- Boot Stirrups (Active Comparator): Participants in this arm will have their feet placed in boot stirrups. Patients will then undergo scheduled vaginal surgery and be asked to complete PROMIS questionnaires before and after surgery.
  Interventions: Procedure: Vaginal Surgery

INTERVENTIONS:
Procedure: Vaginal Surgery — Patients will undergo elective surgery on vagina or bladder

SUMMARY:
The primary objective is to assess the impact of patient positioning using the candy cane stirrups as compared to boot stirrups on physical functioning outcomes at 6 weeks post-op

DETAILED DESCRIPTION:
Patient positioning is an important component of vaginal surgery allowing the surgeon access to the vagina while minimizing patient discomfort and neurological injury. The data on appropriate patient positioning for gynecological vaginal surgery is limited with most providers basing the choice between candy cane and boot stirrups on personal preference. This study has the following aims:

* Aim 1: To perform a randomized controlled trial comparing candy cane stirrups to boot stirrups in patients undergoing vaginal surgery with the primary outcome of change in physical function at 6 weeks post-op as measured by the Patient-Reported Outcomes Measurement and Information System (PROMIS®) 20-Item Physical Functioning Short-Form.
* Aim 2: The investigators aim to measure the angles at the level of hip, knee and foot joints during the surgery in both the candy cane and boot stirrups to assess any association between angles and physical function

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* English speaking
* Scheduled to undergo vaginal or urological surgery with University of Louisville Urogynecology physicians

Exclusion Criteria:

* Immobile or wheelchair bound
* Pre-existing neurological condition limiting physical function
* Age < 18 years
* Patient's with dementia or unable to give informed consent
* Non-English speaking
* Unwilling to follow up in 6 weeks
* Patient's undergoing laparoscopic, robotic or abdominal surgery or surgery through a combined approach
* Patients undergoing surgery under local anesthesia
* Patients who will be awake during positioning

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female gender identity
Enrollment: 155 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement and Information System(PROMIS) Physical Function Scale | preop and 6 weeks post op
  Patients will complete the 20 point Physical Function short form. The minimum score for this scale is 20 and maximum score is 100. A higher score is associated with a better physical function outcome.

SECONDARY OUTCOMES:
Angles of positioning | Intra-operative
  angles at the level of hip, knee and foot joints during the surgery in both the candy cane and boot stirrups to assess any association between angles and physical function

CONTACTS AND LOCATIONS:
Overall Officials: Sean L Francis, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Physicians, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fleisch MC, Bremerich D, Schulte-Mattler W, Tannen A, Teichmann AT, Bader W, Balzer K, Renner SP, Romer T, Roth S, Schutz F, Thill M, Tinneberg H, Zarras K. The Prevention of Positioning Injuries during Gynecologic Operations. Guideline of DGGG (S1-Level, AWMF Registry No. 015/077, February 2015). Geburtshilfe Frauenheilkd. 2015 Aug;75(8):792-807. doi: 10.1055/s-0035-1557776. PMID 26365999
- [Background] Bohrer JC, Walters MD, Park A, Polston D, Barber MD. Pelvic nerve injury following gynecologic surgery: a prospective cohort study. Am J Obstet Gynecol. 2009 Nov;201(5):531.e1-7. doi: 10.1016/j.ajog.2009.07.023. Epub 2009 Sep 17. PMID 19761997
- [Background] Gumus E, Kendirci M, Horasanli K, Tanriverdi O, Gidemez G, Miroglu C. Neurapraxic complications in operations performed in the lithotomy position. World J Urol. 2002 May;20(1):68-71. doi: 10.1007/s00345-001-0241-4. PMID 12088195
- [Background] Cardosi RJ, Cox CS, Hoffman MS. Postoperative neuropathies after major pelvic surgery. Obstet Gynecol. 2002 Aug;100(2):240-4. doi: 10.1016/s0029-7844(02)02052-5. PMID 12151144
- [Background] Litwiller JP, Wells RE Jr, Halliwill JR, Carmichael SW, Warner MA. Effect of lithotomy positions on strain of the obturator and lateral femoral cutaneous nerves. Clin Anat. 2004 Jan;17(1):45-9. doi: 10.1002/ca.10168. PMID 14695587
- [Background] Power H. Patient positioning outcomes for women undergoing gynaecological surgeries. Can Oper Room Nurs J. 2002 Sep;20(3):7-10, 27-30. PMID 12271555
- [Background] Sung VW, Wohlrab KJ, Madsen A, Raker C. Patient-reported goal attainment and comprehensive functioning outcomes after surgery compared with pessary for pelvic organ prolapse. Am J Obstet Gynecol. 2016 Nov;215(5):659.e1-659.e7. doi: 10.1016/j.ajog.2016.06.013. Epub 2016 Jun 16. PMID 27319365
- [Derived] Gupta A, Meriwether K, Tuller M, Sekula M, Gaskins J, Stewart JR, Hobson D, Cardenas-Trowers O, Francis S. Candy Cane Compared With Boot Stirrups in Vaginal Surgery: A Randomized Controlled Trial. Obstet Gynecol. 2020 Aug;136(2):333-341. doi: 10.1097/AOG.0000000000003954. PMID 32649498